CLINICAL TRIAL: NCT00891436
Title: Comparison of the Effect of Fluticasone Furoate Nasal Spray Versus Placebo on Allergic Mediators in the Tears of Subjects With Tree or Grass Pollen Allergy
Brief Title: Study of the Effect of Fluticasone Furoate Nasal Spray on Spring Allergy Eye Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, James Moy, MD, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RUMCgsk 113002
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Results first posted 2012-10-18 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Allergic Conjunctivitis to Tree Pollen or Grass Pollen
MeSH Terms: interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo nasal spray (Placebo Comparator)
  Interventions: Drug: Placebo nasal spray
- Fluticasone furoate nasal spray (Active Comparator)
  Interventions: Drug: Fluticasone furoate nasal spray

INTERVENTIONS:
Drug: Fluticasone furoate nasal spray — 2 sprays each nostril every morning for 2 weeks
  Other Names: Veramyst
  Arms: Fluticasone furoate nasal spray
Drug: Placebo nasal spray — 2 sprays each nostril every morning for 2 weeks
  Arms: Placebo nasal spray

SUMMARY:
Rationale and objectives:

Fluticasone furoate nasal spray (Veramyst) has been shown to improve ocular symptoms when used for the treatment of seasonal allergic rhinitis during the ragweed pollen season. Although this is the only published report of an intranasal corticosteroid shown to effectively treat ocular symptoms, the mechanism has not been delineated. Furthermore, the tears of patients with allergic conjunctivitis are known to have increased concentrations of cytokines and allergic mediators.

The objective of this study is to determine if the positive effects of Veramyst nasal spray on ocular symptoms is via the inhibition of allergic mediators in the eyes. The investigators will conduct a double blind placebo controlled trial to determine if Veramyst nasal spray decreases the amount of allergic mediators in the tears of subjects randomized to Veramyst nasal spray versus placebo. The investigators will also compare the subjects' symptoms to the amount of allergic mediators detected in their tears.

ELIGIBILITY:
Inclusion Criteria:

* a documented history of allergic rhinitis and conjunctivitis due to tree pollen and / or grass pollen for two allergy seasons
* positive skin prick test to tree and / or grass

Exclusion Criteria:

* glaucoma
* cataracts
* acute or chronic sinusitis
* asthma
* chronic obstructive pulmonary disease
* physical nasal obstruction
* pregnant or breastfeeding
* have had a viral or bacterial infections within 2 weeks of the study commencement
* receiving allergen immunotherapy
* have used inhaled corticosteroids within 14 days prior to the study
* have used systemic corticosteroids within 30 days of the study
* travel outside of the geographic area during the 2 week study period
* use of contact lenses during the study period
* use of artificial tears during the study period
* use of eyewash irrigation during the study period
* use of lubricants during the study period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-04; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Moy, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited during the spring pollen season of 2009 at a large urban medcial center's allergy clinic.
Pre-assignment Details: There was no run in period. All 20 participants that enrolled in this study were included in the trial.
Groups:
- Fluticasone Furoate Nasal Spray: Fluticasone furoate nasal spray : 2 sprays each nostril every morning for 2 weeks
- Placebo Nasal Spray: Placebo nasal spray : 2 sprays each nostril every morning for 2 weeks
Period: Overall Study
Arm/Group | Fluticasone Furoate Nasal Spray | Placebo Nasal Spray
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluticasone Furoate Nasal Spray | Placebo Nasal Spray | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32 (7.3) | 29 (8.0) | 30 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Eosinophilic Cationic Protein (ECP) Levels
Description: Tear samples from the participants eyes were collect and were to be used for measuring esinophilic cationic prtein, but this was not measured because the volume of tears were to low.
Time Frame: Samples taken at initial visit & 2 week follow-up
Population: Tear samples from the participants eyes were collect and were to be used for measuring esinophilic cationic prtein, but this was not measured because the volume of tears were to low.
Arm/Group | Fluticasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Histamine Content in the Tears Was Measured.
Description: Tear samples were assayed for histamine by ELISA
Time Frame: Samples taken at initial visit & 2 week follow-up
Population: All participants had tears measured for histamine.
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Fluticasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 10 | 10
ng/ml | 5.4 (0.9) | 5.1 (0.6)
Statistical Analysis 1: Comparison: Fluticasone Furoate Nasal Spray vs Placebo Nasal Spray; paired t-test was used for the data analysis; Test type: Superiority or Other; p > 0.1, t-test, 2 sided; Mean Difference (Final Values) = 2.0, Standard Error of Mean 0.5
Statistical Analysis 2: Comparison: Fluticasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Non-Inferiority or Equivalence — t-test showed no different between the 2 groups; p > 0.1, t-test, 2 sided; Mean Difference (Final Values) = 2.0, Standard Error of Mean 0.5

ADVERSE EVENTS:
Arm/Group | Fluticasone Furoate Nasal Spray | Placebo Nasal Spray
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor has the right to review the results prior to publication of the results. But no embargo or time limit was given.